CLINICAL TRIAL: NCT06401928
Title: Electrical Brain Stimulation for Improving Mental Health and Cognitive Functioning in Patients With Multiple Sclerosis
Brief Title: Electrical Brain Stimulation for Treatment of Secondary Symptoms in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Mohaghegh Ardabili University (Unknown)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, The National Brain Mapping Laboratory (NBML)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPM-MAU
Record Dates: First submitted 2024-05-01; First posted 2024-05-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active tDCS group (Active Comparator): The patients in this group receive 10 daily sessions of 1.5-mA transcranial direct current stimulation (tDCS) targeting the left lateral prefrontal cortex and right orbitofrontal cortex with anodal and cathodal stimulation respectively.
  Interventions: Device: transcranial direct current stimulation
- tDCS with cognitive rehabilitation group (Experimental): The patients in this group receive 10 daily sessions of 1.5-mA transcranial direct current stimulation (tDCS) followed by a 30-minute cognitive training intervention.
  Interventions: Device: transcranial direct current stimulation combined with cognitive training
- sham tDCS group (Sham Comparator): The patients in this group receive 10 daily sessions of 1.5-mA sham transcranial direct current stimulation (tDCS).
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Patients will receive 10 sessions of either 1.5 mA electrical stimulation for 20 minutes each day over 10 consecutive days.
  Arms: active tDCS group
Device: transcranial direct current stimulation combined with cognitive training — Patients will receive 10 sessions of 20 minutes of 1.5 mA electrical stimulation on 10 consecutive days. Each session is followed by 30 minutes cognitive training in which patients conduct several computerized cognitive tests.
  Arms: tDCS with cognitive rehabilitation group
Device: transcranial direct current stimulation — Patients will receive 10 sessions of sham (placebo) electrical stimulation for 20 minutes each day over 10 consecutive days.
  Arms: sham tDCS group

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune disease associated with physical disability, psychological impairment, and cognitive dysfunction. As a result, the disease burden is high, and treatment options are limited. In this randomized, double-blind study, the investigators planned to use repeated electrical stimulation and assess mental health-related variables (e.g., quality of life, sleep, psychological distress) and cognitive dysfunction in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of MS according to the diagnostic criteria for multiple sclerosis: 2010 Revisions to the McDonald criteria (Polman et al., 2011), certified by a professional neurologist
2. being 25-55 years old
3. providing written informed consent
4. If female, a negative urine pregnancy test
5. stable medication regime especially the classical neuroleptics and all CNS-activating medications, if taken, 4-6 weeks before the experiment and during the experiment
6. right handed

Exclusion Criteria:

1. smoker
2. pregnancy
3. alcohol or substance dependence
4. history of seizure
5. history of other neurological disorders than MS
6. history of head injury
7. presence of ferromagnetic objects in the body that are contraindicated for brain stimulation of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Multiple Sclerosis Impact Scale (MSIS-29) | up to 1 day after the intervention
  The MSIS-29 is a questionnaire that comprises of 29 questions. The initial 20 questions are related to the physical impact, whereas the last 9 questions focus on the psychological impact. Each question is rated on a scale of 1 to 5, where 1 indicates "not at all" and 5 indicates "extremely". There are five response options available for the respondents to choose from.
and Depression Anxiety Stress Scale-21 (DASS-21) | up to 1 day after the intervention
  The DASS-21 is a tool used to assess the severity of symptoms related to depression, anxiety, and stress in individuals who have not been diagnosed before. The assessment has three scales, and responses to each are measured on a four-point Likert scale, ranging from 0 to 3.
Mini sleep questionnaire (MSQ) | up to 1 day after the intervention
  The Mini Sleep Questionnaire (MSQ) is used to screen for sleep disturbances in clinical populations. It consists of 10 items, each scored on a seven-point Likert scale ranging from "never" to "always". The questionnaire measures insomnia and oversleeping, with a high score indicating excessive sleepiness and a low score indicating insomnia.

SECONDARY OUTCOMES:
psychomotor speed task | up to 1 day after the intervention
  Performance in the psychomotor speed task (Reaction Time task)
attention / vigilance task | up to 1 day after the intervention
  Performance in the attention / vigilance task (Rapid Visual Information Processing task)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Sclerosis Association of Guilan, Rasht, Giulan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zakibakhsh N, Basharpoor S, Ghalyanchi Langroodi H, Narimani M, Nitsche MA, Salehinejad MA. Repeated prefrontal tDCS for improving mental health and cognitive deficits in multiple sclerosis: a randomized, double-blind, parallel-group study. J Transl Med. 2024 Sep 13;22(1):843. doi: 10.1186/s12967-024-05638-1. PMID 39272101